CLINICAL TRIAL: NCT03136042
Title: A Randomized Crossover Study of Sputum Induction by Physiotherapy and Hypertonic Saline Techniques in Asthmatic Children.
Brief Title: Sputum Induction by Physiotherapy and Hypertonic Saline Techniques in Asthmatic Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Universidade Cidade de Sao Paulo (Other)
Responsible Party: Principal Investigator, Beatriz Mangueira Saraiva Romanholo, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UNICID
Record Dates: First submitted 2017-04-27; First posted 2017-05-02 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Physical Therapy Modalities; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Patients were randomized in first visits into crossover techniques: (i) hypertonic saline (3%) - HS technique; (ii) physiotherapy techniques (oscillatory positive expiratory pressure, forced expiration and acceleration of expiratory flow) - P technique; (iii) hypertonic saline + physiotherapy techniques - HSP technique. All children attended three visits and 90 samples were collected. All patients underwent induced sputum and pulmonary function before and after bronchodilator.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- physiotherapists maneuvers (Experimental): physiotherapy techniques
  Interventions: Other: physiotherapy techniques
- hypertonic saline 3% (Active Comparator): four nebulizations with 3% hypertonic saline.
  Interventions: Other: hypertonic saline 3%
- saline + physiotherapy maneuvers (Active Comparator): 1 nebulizations + physiotherapy techniques
  Interventions: Other: saline + physiotherapy maneuvers

INTERVENTIONS:
Other: physiotherapy techniques — oscillating positive expiratory pressure during nonstop 5 minutes. After that more five minutes to a forced expiratory technique
  Arms: physiotherapists maneuvers
Other: hypertonic saline 3% — four nebulizations with 3% hypertonic saline, the aerosol was generated by an ultrasonic nebulizer
  Arms: hypertonic saline 3%
Other: saline + physiotherapy maneuvers — sputum induction by hypertonic saline at 3% for seven minutes. And more five minutes under physiotherapists maneuvers
  Arms: saline + physiotherapy maneuvers

SUMMARY:
This study evaluated whether physiotherapy is efficient in sputum induction and in evaluation of pulmonary inflammation in asthmatic children.

DETAILED DESCRIPTION:
The hypertonic saline is a traditional technique to collect induced sputum, it´s safe and viable in asthmatic children, as well as the technique of sputum induction and processing has been standardized for schoolchildren.

Sometimes researchers have difficulties to obtain induced sputum in stable patients and it´s possible to use physiotherapy maneuvers to induced sputum. The manouvers are safe for adult and children asthmatics stable.

This study aimed to evaluate the effectiveness to collect induced sputum by physiotherapy maneuvers.

ELIGIBILITY:
Inclusion Criteria:

* Asthmathic children used inhaled corticosteroids not associated with long-acting beta2-agonist.

Exclusion Criteria:

* Asthmathic children to diagnose with other chronic pulmonary pathologies (cystic fibrosis, ciliary dyskinesia, bronchiolitis obliterans, and bronchopulmonary dysplasia) before study, no significant pulmonary pathologies, incapacity to realize pulmonary function and insufficient sample.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2016-01-15 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2018-07-05 (Actual)

PRIMARY OUTCOMES:
Sputum induction by physiotherapists maneuvers | 3 days
  children were seated in a position where the thorax was inclined forwards by 45°, they were instructed to perform calm and long exhalations by oscillating positive expiratory pressure (OPEP) during nonstop 5 minutes holding a Flutter® (Scandipharm, Birmingham, AL, EUA). After that, children were positioned in supine zero degree and underwent for more five minutes to a forced exhalation with the open mouth/glottis (huffing) associated to acceleration by forced expiratory technique (FET), performed by the therapist by positioning a hand on xiphoid process and the other in the manubrium sternum.

SECONDARY OUTCOMES:
Sputum induction by hypertonic saline 3% | 3 days
  children received until four nebulizations with 3% hypertonic saline, the aerosol was generated by an ultrasonic nebulizer (Ultraneb 99; DeVilbiss, Somerset, PA) each challenge was monitored with PEF between nebulizations.

OTHER OUTCOMES:
Sputum induction by hypertonic saline 3% associated with physiotherapists maneuvers | 3 days
  Firstly, children underwent sputum induction by hypertonic saline at 3% for seven minutes. Second, they underwent five minutes OPEP and then five minutes of huffing and FET, as described above.

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz s Romanholo, Dr, Principal Investigator — Universidade Cidade de Sao Paulo
Locations (1):
- Children's Institute of the Clinical Hospital of University of Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Felicio-Junior EL, Barnabe V, de Almeida FM, Avona MD, de Genaro IS, Kurdejak A, Eller MCN, Verganid KP, Rodrigues JC, Tiberio IFLC, Martins MA, Saraiva-Romanholo BM. Randomized trial of physiotherapy and hypertonic saline techniques for sputum induction in asthmatic children and adolescents. Clinics (Sao Paulo). 2020 Jan 24;75:e1512. doi: 10.6061/clinics/2020/e1512. eCollection 2020. PMID 31994616
- Available data/document: references — https://www.ncbi.nlm.nih.gov/pubmed/ — GINA. Global Strategy for Asthma Management and Prevention NHLBI/WHO Workshop Report 2012. 2012 ISAAC. Worldwide variations in the prevalence of asthma symptoms: the International Study of Asthma and Allergies in Childhood (ISAAC). Eur Respir J 1998; 12:315-335 Solé D, Wandalsen GF, Camelo-Nunes IC, et al. Prevalence of symptoms of asthma, rhinitis, and atopic eczema among Brazilian children and adolescents identified by the International Study of Asthma and Allergies in Childhood (ISAAC) - Phase 3. J Pediatr (Rio J) 2006; 82:341-346 Barnabé V, Saraiva B, Stelmach R, et al. Chest physiotherapy does not induce bronchospasm in stable asthma. Physiotherapy 2003; 89:714-719 ATS. Standardization of Spirometry - American Thoracic Society. Am J Respir Crit Care Med 1995; 152:1107-1136 Saraiva-Romanholo BM, Barnabe V, Carvalho AL, et al. Comparison of three methods for differential cell count in induced sputum. Chest 2003; 124:1060-1066